CLINICAL TRIAL: NCT03159676
Title: Proton-Based Stereotactic Ablative Body Radiotherapy (SABR) for Select Patients With Clinically Localized Prostate Cancer.
Brief Title: Proton-Based Stereotactic Ablative Body Radiotherapy for Prostate Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bradley (Brad) Stish, Principal Investigator, Mayo Clinic
Other Study IDs: 17-000680; ROR1752 (Other: Mayo Clinic); NCI-2024-01752 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Radiation therapy; Radiotherapy; Proton; Proton beam; Stereotactic ablative body radiotherapy; Stereotactic body radiotherapy; SABR; SBRT; Localized; Low risk; Intermediate risk
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Proton Therapy; Radiotherapy; Radiosurgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Radiation: Proton beam — Proton beam
  Other Names: Radiation therapy; Radiotherapy; Stereotactic ablative body radiotherapy; Stereotactic body radiotherapy; SABR; SBRT

SUMMARY:
Stereotactic ablative body radiotherapy (SABR), or stereotactic body radiotherapy (SBRT), is a specialized form of radiotherapy used to treat prostate cancer with five treatments over two weeks, compared with a conventional eight-week or longer treatment course. The purpose of this trial is to investigate the effect that proton-based SABR has on quality-of-life in patients with localized prostate cancer. The evaluation and treatment will otherwise follow standard of care, and is not considered investigational.

DETAILED DESCRIPTION:
Patients with low-risk or intermediate-risk, clinically localized prostate cancer will be evaluated according to standard of care medical practices. The evaluation includes history and examination, prostate-specific antigen (PSA) blood testing, and review of the prior prostate biopsy pathology report; radiology scans (for example, computed tomography [CT], magnetic resonance imaging [MRI], radionuclide bone scan) may be done also; recently completed testing may not need to be repeated. Small markers will be placed in the prostate to guide the proton beam stereotactic ablative body radiotherapy (SABR) treatments, and a hydrogel spacer may also be placed between the prostate and the rectum to push the rectum away from the prostate; the hydrogel spacer will dissolve a few months later. Participants will receive five (5) proton SABR treatments over a two (2) week time period. The study will have participants complete a quality-of life questionnaire and be evaluated for side-effects before starting SABR, at the end of SABR, at three (3), six (6) and 12 months after SABR, and then yearly for five (5) years. Evaluation of the cancer status will follow standard of care practices for at least ten (10) years.

ELIGIBILITY:
Inclusion Criteria:

* Male, age ≥ 18 years.
* Histological confirmation of adenocarcinoma of prostatic origin.
* AJCC 7th edition clinical T1b-fdiabetes mellitus T2b.
* AJCC clinical staging rules do not include findings from biopsy or imaging.
* Gleason score ≤7 (International Society of Urological Pathologists grades 1-3).
* Serum prostate-specific antigen ≤20 ng/mL.
* Prostate-specific antigen <10 ng/mL, if dutasteride within last 90 days or finasteride within last 30 days.
* Zubrod performance score 0-1.
* Prostate volume <75-cc, determined by ultrasound, computed tomography or magnetic resonance imaging (modality with lesser volume is acceptable).
* If neoadjuvant-concurrent androgen suppression is used, the prostate volume after the start of androgen suppression may be used.
* American Urological Association voiding symptom index ≤15.
* Ability to complete questionnaire(s) by themselves or with assistance.
* Participation in a patient-reported outcomes survey program, inclusive of the Expanded Prostate Index Composite and CTCAE instruments.
* Ability to provide informed written consent.

Exclusion Criteria:

* Radiological- or pathologically-confirmed seminal vesicle invasion, lymph node involvement, or distant metastatic disease.

  * Radiological- or biopsy-confirmed extraprostatic tumor extension without AJCC 7th edition clinical T3a classification remain eligible.
* Prior or anticipated external radiotherapy or brachytherapy, transurethral resection of the prostate, prostatic cryoablation/focused ultrasound/laser therapy, prostatectomy, or prostatic enucleation.
* Prior bilateral orchiectomy, planned long-term (>6 months duration) androgen suppression or peripheral androgen blockade, or chemotherapy or immunotherapy for prostate cancer.
* Prior hemi- or total hip arthroplasty.
* Diabetes mellitus associated with vascular ulcers or wound healing problems, ulcerative colitis, connective tissue disorder, or chronic (≥120 days) warfarin or clotting factor inhibitor (e.g., rivaroxaban) use planned.
* Co-morbid severe concurrent disease which, in the judgment of the investigator, would result in life expectancy <5 years.

  * Patients with a left cardiac ventricular assist device are ineligible.
  * Patients with an implanted medical electronic device (e.g., cardiac pacemaker) remain eligible if device monitoring complies with standard of practice (e.g., Cardiology and Medical Physics evaluation, function checks and during-treatment monitoring).
* Immunocompromised due to HIV positive state.
* Medical or psychiatric conditions that preclude informed decision-making or adherence.
* Prior registration to an Institutional Review Board-approved therapeutic research study that includes proton beam therapy or photon-based radiotherapy (e.g., randomization to proton beam therapy vs. photon-based radiotherapy).

  * Registration to a non-therapeutic (e.g., biomarker, medical physics) only research study is not an exclusion.
* Inability to start radiation per protocol.

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Adult male patients with prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-05-12 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 24 months
  Will be assess by the number of late grade ≥3 Gastrointestinal and Renal and Urinary/Genitourinary adverse event incidents recorded at 24 months after SABR

SECONDARY OUTCOMES:
Biochemical (PSA) failure | 120 months
  Assessed as time from registration until the date prostate-specific antigen value is ≥ prostate-specific antigen nadir + 2.0 ng/mL estimated by the Gray cumulative incidence method.
Quality of life - EPIC | Baseline; 120 months
  Assessed using the Expanded Prostate Index Composite (EPIC). The EPIC consists of 13 questions answered on varying 5-point scales (e.g., Very Poor/Non to Very Good or No Problem to Big Problem). Subdomains for urinary, bowel, and sexual function will be summarized descriptively. Changes across time will be evaluated to assess patient function and quality of life after study treatment.
Overall survival | 120 months
  Overall survival is defined as the length of time participants are alive after the start of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Brad J. Stish, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Proton Beam Therapy Clinical Trials — http://www.mayoclinic.org/departments-centers/proton-beam-therapy-program/sections/clinical-trials/rsc-20185494